CLINICAL TRIAL: NCT03543449
Title: Predictability of Preoperative Hemoglobin A1c in Diabetic Patients Underwent Off-Pump Coronary Artery Bypass Surgery: A Retrospective Study.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0221
Record Dates: First submitted 2018-05-20; First posted 2018-06-01 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease, Diabetes
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus | interventions — Coronary Artery Bypass, Off-Pump; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Off-Pump Coronary Artery Bypass (OPCAB) surgery — Off-Pump Coronary Artery Bypass (OPCAB) surgery. This study is retrospective study

SUMMARY:
The aim of this study is to evaluate evaluated the impact of preoperative HbA1c in diabetic patients on perioperative glycemic variability and outcome after off-pump coronary artery bypass (OPCAB).

The medical records of patients who had a preoperative diagnosis of diabetes and underwent OPCAB from 2005 to 2017 will be reviewed. Patients are divided by HbA1c levels (<7.0% or ≥7.0%). Glycemic variability during surgery and up to 24 hours after surgery is assessed by the coefficient of variation. The primary outcome is defined as a composite of postoperative permanent stroke, prolonged ventilation, deep sternal wound infection, renal failure, reoperation, mortality according to the definition of STS (Society of Thoracic Surgery) version 2.81 adult cardiac surgery database. If one or more of the above five morbidity or mortality occur, it is assumed that composite morbidity/mortality had occurred. We compare postoperative complications, mortality and perioperative glycemic variability between patients with HbA1c ≥7.0% and <7.0%, and examined the effects of perioperative glycemic control on postoperative morbidity and mortality (composite morbidity/mortality).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of preoperative diabetes mellitus and with available results of HbA1c test within 3 months before surgery.
* Patients who aged 20 to 89 years

Exclusion Criteria:

* Patient who had a history of previous coronary artery bypass surgery
* Patients whose surgery plan changed to cardiopulmonary bypass during surgery.

Ages: 20 Years to 89 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a history of preoperative diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 703 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Permanent stroke | during the hospitalization for surgery (up to 30 days)
  postoperative stroke (i.e., any confirmed neurological deficit of abrupt onset caused by a disturbance in blood supply to the brain that did not resolve within 24 hours.)
Incidence of Renal failure | during the hospitalization for surgery (up to 30 days)
  1. Increase in serum creatinine level 3.0 x greater than baseline, or serum creatinine level ≥ 4 mg/dL. The acute rise must be at least 0.5 mg/dl.
  2. A new requirement for dialysis postoperatively.
Incidence of Prolonged ventilation | during the hospitalization for surgery (up to 30 days)
  Prolonged post-operative pulmonary ventilation > 24.0 hours. The hours of postoperative ventilation time include OR exit until extubation, plus any additional hours following reintubation.
Incidence of Deep sternal wound infection | during the hospitalization for surgery (up to 30 days)
  Deep sternal wound infection or mediastinitis including muscle layer according to CDC definition
Incidence of Re-operation for any reason | during the hospitalization for surgery (up to 30 days)
  reoperation for bleeding/tamponade, valvular dysfunction, graft occlusion, other cardiac reason, or non-cardiac reason
Operative mortality | during the hospitalization for surgery (up to 30 days)
  all deaths, regardless of cause

SECONDARY OUTCOMES:
Perioperative Coefficient of variation of glucose | During surgery and up to the first 24 hours after surgery
  the standard deviation divided by the average of blood glucose concentration during surgery and first 24 hours after surgery
Incidence of Perioperative Coefficient of variation of glucose | During surgery and up to the first 24 hours after surgery
  the standard deviation of blood glucose concentration during surgery and first 24 hours after surgery
Perioperative mean glucose | During surgery and up to the first 24 hours after surgery
  average of blood glucose concentration during surgery and first 24 hours after surgery
Perioperative time-weighted average glucose | During surgery and up to the first 24 hours after surgery
  time-weighted average of blood glucose concentration during surgery and first 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology & Pain Medicine, Yonsei university college of medicine, Seoul, South Korea